CLINICAL TRIAL: NCT03882268
Title: A Feasibility Study of Integrating Maternal, Infant and Young Child Nutrition (MIYCN) Counseling Services in Urban Maternal, Neonatal and Child Health (MNCH) Services in Bangladesh: A Quasi-experimental Evaluation
Brief Title: Integrating MIYCN Counseling in Urban Health Services
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: International Food Policy Research Institute (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: InternationalFPRI
Record Dates: First submitted 2019-03-12; First posted 2019-03-20 (Actual); Last update posted 2023-09-26 (Actual); Status verified 2022-02

CONDITIONS: Maternal Nutrition
Keywords: Urban; Maternal Nutrition; Nutrition Counseling; Behavior change; Infant and young child feeding

STUDY DESIGN:
Intervention Model Description: 8 NGO-run urban health facilities in Dhaka will receive intensified MIYCN interventions, while another 8 NGO-run urban health facilities will serve as a comparison group. No randomization will take place. No randomization will take place. Health workers and clients at these facilities will be participants in the study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- MIYCN interventions (Experimental): 8 facilities run by 2 NGOs that will receive intensified MIYCN interventions.
  Interventions: Behavioral: MIYCN interventions
- Comparison facilities (No Intervention): 8 facilities run by 2 other NGOs, which will not receive any standardized MIYCN interventions.

INTERVENTIONS:
Behavioral: MIYCN interventions — 1. Capacity building for health providers and nutrition counselors (training on MIYCN SBCC from A&T).
  2. Dedicated room for MIYCN counseling at health facilities with standardized layouts, displays of government IYCF logo, and other specifications.
  3. Availability of standardized MIYCN-specific BCC materials and job aids.
  4. Standardized MIYCN counseling services (counseling on diet diversity and quantity, IFA and calcium supplementation, weight gain monitoring, exclusive and early initiation of breastfeeding, complementary feeding, and water, sanitation and health) provided by a dedicated MIYCN counselor hired by A&T.
  5. Dedicated community worker hired by A&T to identify and mobilize beneficiaries needing services in the community (via satellite clinic outreach, distribute MIYCN flyers, and provision of MIYCN education via phone or home visits).
  6. Supportive supervision of MIYCN counselors and community workers by program and facility managers, and field supervisors.
  Arms: MIYCN interventions

SUMMARY:
The study will use a quasi-experimental design to examine the feasibility of standardizing MIYCN counseling services in existing health facilities to improve the quality of MIYCN services. The impact of standardized and upgraded services on client utilization, knowledge and behavior will also be measured. 8 NGO-run urban health facilities in Dhaka will receive intensified MIYCN interventions, while another 8 NGO-run urban health facilities will serve as a comparison group. No randomization will take place.

DETAILED DESCRIPTION:
The primary objectives of the proposed evaluation are to answer the following questions:

* Is it feasible to standardize the delivery of MIYCN counseling services in existing urban health facilities?
* Can quality of MIYCN counseling service be improved by upgrading and standardizing existing MIYCN counseling service in urban health facilities?
* What are the impacts of standardized and upgraded MIYCN counseling service on utilization of MIYCN services and knowledge of clients?

The secondary objectives are:

* What are the impacts of standardized and upgraded MIYCN counseling service on behaviors of clients including:

  * Pregnant women: 1) consumption of diversified foods; 2) intake of IFA and calcium supplements during pregnancy
  * Mothers of children <1 y: age-appropriate infant feeding

The study will use a quasi-experimental design, with data collection taking place in three different stages: 1) Baseline data collection to assess comparability of facilities, service quality and client's behaviors, 2) Facility-based endline data collection and 3) Community-based endline survey.

The evaluation was originally intended to be a randomized control trial, covering 20 NGO-run urban health facilities under contract with the Urban Primary Health Care Services Delivery Project (UPHCSDP). 10 of the 20 health facilities were randomized to receive the intervention, while the other 10 facilities would serve as the comparison group. Baseline data collection took place in these 20 facilities in October-November 2019. However, the project did not receive approval from UPHCSDP, and interventions were not implemented at the 10 facilities in the treatment group.

Instead, A&T partnered with 2 other NGOs in Dhaka whose 8 health facilities also provide services in urban areas but are not affiliated with UPHCSDP. These 8 facilities will receive the intervention. Propensity score matching will be used to select 8 of the original 20 facilities under contract with UPHCSDP to serve as the control group.

Baseline data collection in the intervention facilities will take place in February-March 2020. The facility-based end line will take place in May-June 2022, and the community-based endline will take place in June 2022. Data will be collected for the full sample of intervention facilities at baseline (i.e. with the same sample size as at endline), given uncertainty in obtaining government approval to collect endline data from comparison facilities under contract with UPHCSDP. The larger sample from intervention facilities at baseline allows for a shift in evaluation design from quasi-experimental to a pre-post comparison, if the project does not receive government approval.

The study will use mixed data collection methods including: 1) facility assessment; 2) provider survey; 3) case observations (namely ANC visits, child visits [both sick child and immunization], and counseling sessions), 4) client interviews and 5) in-depth interview with Program Managers and Field Supervisors.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women who are visiting the health facilities for ANC visits (at least twice during her pregnancy, around half of clients)
* Mothers with children <12 months of age who are visiting the health facilities for health check-ups or vaccination

Exclusion Criteria:

* Pregnant women with severe illness or complications
* Mothers with severely ill children

Ages: 18 Years to 49 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 4128 (Actual)
Dates: Start 2019-11-15 (Actual); Primary Completion 2022-06-30 (Actual); Study Completion 2022-11-30 (Actual)

PRIMARY OUTCOMES:
Facility readiness for nutrition services | 15-16 months after baseline in a cross-sectional endline survey scheduled for May-June 2022
  Total standardized scores of resources and staffing available to provide nutrition services at the health facility, with higher scores representing higher readiness.
Service provider knowledge on topics related to maternal and child nutrition | 15-16 months after baseline in a cross-sectional endline survey scheduled for May-June 2022
  Total standardized scores of correct answers to questions related to maternal and child nutrition, with higher scores represent higher knowledge.
Quality of nutrition counseling during ANC by health staff | 15-16 months after baseline in a cross-sectional endline survey scheduled for May-June 2022
  Total standardized scores of correct messages on diet diversity and quantity, IFA and calcium supplementation, weight gain monitoring, early initiation of breastfeeding, and water, sanitation and health by health staff during counseling sessions, with higher scores representing higher quality of counseling.
Quality of nutrition counseling during well-child or sick-child visits by health staff | 15-16 months after baseline in a cross-sectional endline survey scheduled for May-June 2022
  Total standardized scores of correct messages on exclusive and early initiation of breastfeeding, complementary feeding, and water, sanitation and health provided by health staff during counseling sessions, with higher scores representing higher quality of counseling.
Pregnant women's/mother's utilization of and satisfaction with MIYCN services | 15-16 months after baseline in a cross-sectional endline survey scheduled for May-June 2022
  Total standardized scores of answers to questions related to utilization of and satisfaction with MIYCN services, with higher scores represent higher utilization and satisfaction.
Pregnant women's/mother's knowledge of MIYCN topics | 16 months after baseline in a cross-sectional endline survey scheduled for June 2022
  Total standardized scores of correct answers to questions related to maternal and child nutrition, with higher scores representing higher knowledge.

SECONDARY OUTCOMES:
Diet diversity among pregnant women | 16 months after baseline in a cross-sectional endline survey scheduled for June 2022
  The proportion of pregnant women who consumed foods from 5 or more food groups on the day preceding the interview.
Maternal consumption of IFA tablets | 16 months after baseline in a cross-sectional endline survey scheduled for June 2022
  The mean number of IFA tablets consumed during pregnancy.
Maternal consumption of calcium tablets | 16 months after baseline in a cross-sectional endline survey scheduled for June 2022
  The mean number of calcium tablets consumed during pregnancy.
Early initiation of breastfeeding | 16 months after baseline in a cross-sectional endline survey scheduled for June 2022
  The proportion of women who initiated breastfeeding within one hour of birth.
Exclusive breastfeeding among children aged 0-5.9 months | 16 months after baseline in a cross-sectional endline survey scheduled for June 2022
  The proportion of infants aged less than 6 months who were exclusively breastfed on the day preceding the interview.
Age-appropriate complementary feeding of children aged 6-11.9 months | 16 months after baseline in a cross-sectional endline survey scheduled for June 2022
  The proportion of children aged 6-11.9 months who received foods from 4 or more food groups and fed the appropriate number of times/meals on the day preceding the interview.

CONTACTS AND LOCATIONS:
Overall Officials: Purnima Menon, PhD, Principal Investigator — IFPRI
Locations (1):
- Data Analysis and Technical Assistance Limited, Dhaka, Bangladesh

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Nguyen PH, Sununtnasuk C, Christopher A, Ash D, Ireen S, Kabir R, Mahmud Z, Ali M, Forissier T, Escobar-DeMarco J, Frongillo EA, Menon P. Strengthening Nutrition Interventions during Antenatal Care Improved Maternal Dietary Diversity and Child Feeding Practices in Urban Bangladesh: Results of a Quasi-Experimental Evaluation Study. J Nutr. 2023 Oct;153(10):3068-3082. doi: 10.1016/j.tjnut.2023.06.023. Epub 2023 Jun 23. PMID 37354978

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2021-10-01): https://cdn.clinicaltrials.gov/large-docs/68/NCT03882268/Prot_SAP_000.pdf
  • Informed Consent Form (2021-08-06): https://cdn.clinicaltrials.gov/large-docs/68/NCT03882268/ICF_001.pdf